CLINICAL TRIAL: NCT04729517
Title: Randomized Multicenter Phase III Efficacy and Safety Study of AI201901 in Allergic Rhinitis Patients (HILARIA)
Brief Title: Efficacy and Safety Study of AI201901 in Allergic Rhinitis Patients
Acronym: HILARIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abdi Ibrahim Ilac San. ve Tic A.S. (Industry)
Collaborators: Istanbul Umraniye Training and Research Hospital (Unknown); Diskapi Yildirim Beyazit Education and Research Hospital (Other Government); Antalya Training and Research Hospital (Other Government); Dokuz Eylul University (Other); Ankara City Hospital Bilkent (Other); Kahramanmaras Sutcu Imam University (Other); Uludag University (Other); Karadeniz Technical University (Other); Kartal Dr. Lütfi Kirdar City Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aİ-2019-01
Record Dates: First submitted 2021-01-20; First posted 2021-01-28 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2022-08

CONDITIONS: Allergic Rhinitis Due to Allergens
Keywords: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — azelastine

STUDY DESIGN:
Intervention Model Description: The first group will receive AI201901 , whereas the second group will receive azelastine hydrochloride. Patients that will receive AI201901 are defined as the test arm and patients that will receive azelastine hydrochloride are defined as the active control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azelastine Hydrochloride (Active Comparator): Patients that will receive azelastine hydrochloride are defined as the active control arm.
  Interventions: Drug: Azelastine Hydrochloride
- AI201901 (Experimental): Patients that will receive AI201901 are defined as the test arm.
  Interventions: Drug: AI201901

INTERVENTIONS:
Drug: AI201901 — Twice daily inhaled AI201901 for 4 weeks
  Arms: AI201901
Drug: Azelastine Hydrochloride — Twice daily inhaled Azelastine Hydrochloride for 4 weeks
  Other Names: Allergodil
  Arms: Azelastine Hydrochloride

SUMMARY:
This is a prospective, national, randomized, multicenter, parallel group, Phase III study that evaluates the effects of AI201901 in Allergic Rhinitis patients, where they will spray twice a day against azelastine into both nostrils during a 28-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed as allergic rhinitis on the basis of medical history, physical examination, and skin prick test, and according to ARIA 2008 criteria
* To be included in seasonal and perennial allergic rhinitis group
* To have a related complaint for at least 2 years
* To be informed about the study and to give consent to participate in the study

Exclusion Criteria:

* Diagnosis of superficial nasal mucosal erosion, moderate nasal mucosal erosion, nasal mucosal ulceration and nasal septum perforation during nasal examination
* Presence of nasal diseases that are likely to affect the accumulation of intranasal drugs, such as acute or chronic sinusitis, rhinitis medicamentosa, clinically significant polyposis or clinically significant nasal structural abnormalities
* Having undergone a nasal or sinus surgery for up to one year before the study
* The use of systemic or topical steroids within the last 15 days prior to inclusion in the study
* The use of antihistamine, chromoline Na within the last 15 days prior to inclusion in the study
* The use of any investigational drug within 30 days prior to Visit 1;
* Known hypersensitivity to components of the products used in the study
* Presence of respiratory infections, which have developed within the two weeks prior to Visit 1
* Diagnosis of COPD
* A history of alcohol or drug addiction treatment within the last 2 years prior to inclusion in the study, or any current addiction on alcohol or drugs,
* Use of alcohol and other drugs (antidepressants) that have a negative effect on reaction time / concurrent use of sedative drugs or other drugs that act on the central nervous system
* Presence of significant lung diseases including asthma. ((Only patients with intermittent asthma who need short-acting inhaled bronchodilators (no more than twice a week) and do not wake up at night due to asthma are suitable for inclusion)).
* Presence of chronic obstructive sleep-apnea syndrome (clinical diagnosis)
* Presence of any surgical or medical condition, which, according to the opinion of the responsible researcher, could significantly alter the absorption, distribution, metabolism, or excretion of the investigational product, or could significantly affect the patient's ability to complete this study
* Presence of symptoms in the medical history in relation to glaucoma, cataract, ocular herpes simplex, conjunctivitis, or other ocular infections
* Presence of medical history in relation to active or latent tuberculosis
* Presence or risk of exposure to chickenpox or measles within the last 30 days
* Presence of untreated fungi, bacteria or systemic viral infection within the last 30 days
* Being pregnant or breastfeeding
* Women of reproductive age who do not use a medically valid contraceptive method
* Presence of cystic fibrosis
* Presence of primary ciliary dyskinesia
* Use of intranasal or systemic first-generation antihistamines, leukotriene receptor antagonists or other nasal decongestants during the study
* Use of any ophthalmic steroid or nasal, inhaled or systemic steroid during the study
* Use of another clinical research product during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score | 28 days
  Achieve a statistically significant improvement in the symptoms of allergic rhinitis via Total Nasal Symptom Score (TNSS).

SECONDARY OUTCOMES:
TNNSS; Total non nasal symptom score | 28 days
  In non-nasal symptom scores (TNNSS), AI201901 is similar compared to azelastine
The rhinoconjunctivitis quality of life scale (RQLQ) | 28 days
  The rhinoconjunctivitis quality of life scale (RQLQ) indicates that AI201901 is similar compared to azelastine
Odor Visual Analogue Score (VAS) | 28 days
  In Odor Visual Analogue Score (VAS) results, AI201901 is better than azelastine
Inspiratory peak flow meter (PNIF) | 28 days
  Inspiratory peak flow meter (PNIF) results show that AI201901 is similar compared to azelastine
Connecticut butanol odor threshold test | 28 days
  Connecticut butanol odor threshold tests show that AI201901 is similar compared to azelastine
Rhinoscopic Assessment Scale | 28 days
  Results of the Rhinoscopic Assessment Scale show that AI201901 is better than azelastine
Safety of AI201901 | 28 days
  Demonstration of the safety of AI201901 by comparing the number of participants with treatment-related adverse events in each arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)